CLINICAL TRIAL: NCT04706949
Title: A Prospective, Single Center, Single Arm, Phase II Clinical Trial of Pyrotinib Combined With Pemetrexed Plus Carboplatin in the First-line Treatment of Patients With HER2 Mutant or Amplified Recurrent / Metastatic Non-small Cell Lung Cancer
Brief Title: Pyrotinib Combined With Pemetrexed Plus Carboplatin in the First-line Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jialei Wang, Principal Investigator, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BLTN-HER2-001
Record Dates: First submitted 2020-12-28; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Lung Cancer, Non-small Cell
Keywords: Lung Cancer, Non-small Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib combined with pemetrexed plus carboplatin (Experimental)
  Interventions: Drug: Pyrotinib combined with pemetrexed plus carboplatin

INTERVENTIONS:
Drug: Pyrotinib combined with pemetrexed plus carboplatin — 1. Pyrotinib: oral administration within 30 minutes after breakfast, 400mg / day, continuous administration for 21 days as a cycle; each continuous pause time and the cumulative pause time of each cycle should not exceed 14 days. It is allowed to suspend the drug for many times due to adverse events.
  2. Pemetrexed: the recommended dosage is 500mg / m2, once every three weeks. 3) Carboplatin: the dosage was determined according to Calvert formula, in which AUC was 5mg / ml / min.

SUMMARY:
A prospective, single center, single arm, phase II clinical trial of Pyrotinib combined with pemetrexed plus carboplatin in the first-line treatment of patients with HER2 mutant or amplified recurrent / metastatic non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Aged≥18 and <75 years.
* Histologically or cytologic confirmed Non-small cell lung cancer, Phase IIIB or IV according to UICC 2017.
* ECOG performance status of 0 to 1.
* Life expectancy of more than 3 months.
* Confirmed HER2 mutation and amplification by Central Laboratory. Direct sequencing (RT-PCR or ARMS-PCR) or second generation sequencing (NGS) was used for HER2 mutation, and fluorescence in situ hybridization (FISH) or ngs was used for HER2 amplification;
* At least one RECIST 1.1 defined measurable lesions.
* Patients who had not received systemic treatment for advanced / metastatic NSCLC in the past but had disease progression more than 12 months after receiving neoadjuvant therapy or the last use of adjuvant therapy could be enrolled.
* Required laboratory values including following parameters:ANC≥1.5×109/L,Platelet count≥90×109/L,Hemoglobin≥90 g/L;Total bilirubin:≤ 1.5×upper limit of normal, ULN, ALT and AST≤ 2.0×ULN; BUN and Cr: ≤1.5 x ULN;creatine clearance rate: ≥ 50 mL/min, LVEF: ≥ 50%; QTcF:< 470 ms for female and < 450 ms for male.
* Signed informed consent.

Exclusion Criteria:

* Previous therapy with other HER2 inhibitors.
* Inability to swallow、chronic diarrhea and intestinal obstruction that affect the drug taking and absorption.
* There is unstable third space effusion (such as large amount of pleural effusion and ascites).
* Received radiotherapy, chemotherapy, surgery or other targeted therapy for non-small cell lung adenocarcinoma within 4 weeks before taking the study drug for the first time.
* Persistence of clinically relevant therapy related toxicities from previous therapy (greater than Common Terminology Criteria for Adverse Event(CTCAE) 4.0 grade 1).
* Patients with active brain metastasis (without medical control), cancerous meningitis, spinal cord compression, or diseases of brain or pia mater found by CT or MRI examination during screening (patients with brain metastasis who had completed treatment or stable symptoms within 28 days before taking the study drug for the first time can be enrolled, but they need to be confirmed as having no symptoms of cerebral hemorrhage by MRI, CT or venography evaluation).
* Participated in other drug clinical trials within the past 4 weeks before start of therapy.
* Other malignant tumors in the past 5 years, excluding cervical carcinoma in situ, basal cell carcinoma of skin or squamous cell carcinoma of skin.
* At the same time receive any other anti-tumor treatment, such as immune agents and anti angiogenesis inhibitors.
* Those with allergic constitution or known allergic history to the drug components of the scheme.
* Active infection(judged by the researcher).
* Subjects had any heart disease, including: (1) angina; (2) requiring medication or clinically significant arrhythmia; (3) myocardial infarction; (4) heart failure; (5) Any heart diseases judged by investigator as unsuitable to participate in the trial.
* Female patients who are pregnancy, lactation or women who are of childbearing potential tested positive in baseline pregnancy test.
* According to the judgment of the researchers, there are concomitant diseases (such as uncontrolled hypertension, diabetes, thyroid disease, etc.) that seriously endanger the safety of patients or affect the completion of the study.
* Known history of neurological or psychiatric disease, including epilepsy or dementia.

Any of the other conditions of which researchers believe that the patient is not fit to take part in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | from the first cycle of treatment (day one) to two month after the last cycle (each cycle is 21 days)]
  progression free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No